CLINICAL TRIAL: NCT06371326
Title: A Randomized, Double-blind, Placebo-controlled, Multiple-ascending-dose Phase Ic Study Evaluating the Safety, Tolerability, and Pharmacokinetics of ZT002 Injection in Participants With Overweight or Obesity
Brief Title: A Study of ZT002 Injection in Participants With Overweight or Obesity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing QL Biopharmaceutical Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BJQLZT002004
Record Dates: First submitted 2024-04-10; First posted 2024-04-17 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Overweight or Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ZT002 Injection (Experimental): Participants will be randomized to receive ZT002 injection in 1of 2 dose cohorts.
  Interventions: Drug: ZT002 Injection
- ZT002 Placebo (Placebo Comparator): Participants will be randomized to receive same volume Placebo in 1 of 2 dose cohorts.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ZT002 Injection — Participants will receive ZT002 by subcutaneous (SC) injection.
  Arms: ZT002 Injection
Drug: Placebo — Participants will receive Placebo by subcutaneous (SC) injection.
  Arms: ZT002 Placebo

SUMMARY:
This study will comprise a randomized, double-blind, placebo-controlled, multiple-ascending-dose, safety, tolerability, and pharmacokinetics study of ZT002 in participants with Overweight or Obesity.

ELIGIBILITY:
Inclusion Criteria:

* 1. Males and females aged 18 to 50 years (inclusive, based on age at the time of signing the informed consent form);

  2. BMI ≥ 24 kg/m2 and < 28 kg/m2 with at least one of the following concomitant disease (pre-diabetes [except for type 1 or type 2 diabetes], hypertension, hyperlipidemia, fatty liver, obstructive sleep apnoea syndrome, weight-bearing joint pain, etc., see Appendices I and II) or BMI ≥ 28 kg/m2 and ≤ 40 kg/m2 and with or without concomitant disease;

  3. Weight change of no more than 5% (based on self-report) after 3 months of weight control via diet and exercise alone prior to screening, and the formula for calculating weight change is: (highest weight - lowest weight during 3 months of weight control via diet and exercise alone prior to screening) ∕highest weight*100%;

  4. Female subjects are required to adopt abstinence or 2 effective methods of contraception from 1 month prior to screening to 6 months after the last dose, and male subjects are required to adopt abstinence or 2 effective methods of contraception from the first dose to 3 months after the last dose. For male subjects, the effective methods of contraception are as follows: surgical sterilization (e.g., vasectomy) or proper use of condoms, or the female partners use hormonal contraceptives (e.g., contraceptive pills, patches, implantable or injectable) or intrauterine devices (IUDs) or surgical sterilization; for female subjects, the effective methods of contraception are as follows: surgical sterilization (e.g., tubal ligation) or use of IUDs, or male partners properly use condoms or are surgically sterilized, in addition, the female subjects are allowed to use the NMPA-approved hormonal contraceptives (e.g., contraceptive pills, patches, implantable or injectable);

  5. Subjects who have a good understanding of study objectives, be able to communicate well with the investigator, and be able to understand and comply with the requirements set forth for this study.

Exclusion Criteria:

* 1. History of specific allergies (asthma, eczema, etc.) or allergic constitution, or history of allergy to two or more drugs and foods, especially to the investigational drug and its excipients or GLP-1-containing drugs;

  2. Previous diagnosis of obesity associated with endocrine disease or single gene mutation, including but not limited to, hypothalamic obesity, pituitary obesity, hypothyroid obesity, Cushing's syndrome, insulinoma, acromegaly, hypogonadism;

  3. Subjects who have had severe gastrointestinal diseases (e.g., active ulcers) or undergone gastrointestinal surgery (except for appendectomy or cholecystectomy) or have clinically significant abnormalities of gastric emptying (e.g., pyloric obstruction, gastric paralysis) within 6 months prior to screening or have been taking medications that have a direct effect on gastrointestinal motility for a long term, or who are not suitable for participation in the trial as assessed by the investigator;

  4. Prior history of significant cardiovascular disease, defined as:

  a) History of myocardial infarction, coronary angioplasty or bypass grafting, heart valve disease or heart valve repair, clinically significant arrhythmia requiring treatment, unstable angina pectoris, transient ischemic attack, or cerebrovascular accident within 6 months prior to screening; b) New York Heart Association (NYHA) class III or IV congestive cardiac failure;

  5. Uncontrolled hypertension: systolic blood pressure ≥ 160 mmHg and/or diastolic blood pressure ≥ 100 mmHg;

  6. Laboratory test results at screening meet any of the following criteria (one retest is allowed during the screening period if there is any clear reason, and the investigator should document the reason for retest):
  1. Glycosylated hemoglobin (HbA1c) ≥ 6.5% or fasting plasma glucose ≥ 7.0 mmol/L, or two-hour plasma glucose ≥ 11.1 mmol/L on oral glucose tolerance test (OGTT) (at screening, subjects with fasting venous plasma glucose between 6.1 and 6.9 mmol/L need to perform OGTT) (see Appendix I, OGTT Test Method);
  2. Thyroid-stimulating hormone (TSH) > 6.0 mIU/L or < 0.4 mIU/L;
  3. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≥ 3 × ULN or blood total bilirubin ≥ 2 × ULN;
  4. Fasting triglycerides > 5.65 mmol/L;
  5. Blood amylase or blood lipase ≥ 1.5 × ULN;
  6. Calcitonin ≥ 50 ng/L (pg/mL);
  7. Estimated glomerular filtration rate (eGFR) ≤ 60 mL/min/1.73m2, estimated using CKD-EPI formula (see Appendix 3);
  8. Abnormal 12-lead electrocardiogram (ECG): second- or third-degree atrioventricular block, long QT syndrome or QTcF > 450 ms (males) or > 470 ms (females) (see formula in Appendix 4), left or right bundle branch block, pre-excitation syndrome, or other clinically significant arrhythmia (except for sinus arrhythmia);

     7. Previous history of acute and chronic pancreatitis, history of symptomatic gallbladder disease (except for cholecystectomy), history of pancreatic injury, and other high risk factors for pancreatitis;

     8. Previous personal or family history of medullary thyroid carcinoma (MTC) or type 2 multiple endocrine neoplasia syndrome (MEN2);

     9. Prior diagnosis of malignancy (except for cured basal cell skin cancer or cervix carcinoma in situ);

     10. A past history of hypoglycemia or recurrent symptomatic hypoglycemia (more than twice in 6 months);

     11. Infectious disease (which would affect the subject's ability to participate in the trial as judged by the investigator) within 4 weeks prior to screening;

     12. Use of any prescription, over-the-counter, or Chinese herbal medications within 1 month prior to screening or discontinuation less than 5 drug half-lives (whichever is longer);

     13. Use of any of the following medications or therapies within 3 months prior to screening:

  <!-- -->

  1. Any approved or unapproved weight-loss drugs (e.g., liraglutide, semaglutide, beinaglutide, orlistat, lorcaserin, phentermine/topiramate, naltrexone/bupropion) or weight-affecting Chinese herbal medications, supplements, meal replacements;
  2. Use of any hypoglycemic medications (e.g., sodium-glucose cotransporter protein 2 inhibitors [SGLT2i] and glucagon-like peptide-1 receptor agonists [GLP-1RA], metformin, alpha-glucosidase inhibitors);
  3. Use of medications that may cause significant weight gain, including systemic glucocorticoid therapy; tricyclic antidepressants; antipsychotic or antiepileptic drugs (e.g., clomipramine, amitriptyline, mirtazapine, paroxetine, phenelzine, chlorpromazine hydrochloride, clozapine, olanzapine, valproic acid and its derivatives, lithium preparations, thioridazine), for more than 1 week;

     14. Subject who have prior history of bariatric surgery (except for those who have undergone liposuction more than 1 year ago) or who plan to undergo bariatric surgery or use bariatric equipment during the study period;

     15. Subjects who have undergone surgery within 3 months prior to screening, or plan to undergo surgery during the study, and anyone who has undergone surgery that affects drug absorption, distribution, metabolism, or excretion;

     16. Subjects who have participated in other clinical trials and received drug therapies or medical device interventions within 3 months prior to screening;

     17. Subjects who have been vaccinated within 1 month prior to screening or plan to be vaccinated during the trial;

     18. Donation or loss of blood ≥ 400 mL, or blood transfusion within 3 months prior to screening;

     19. Subjects who cannot tolerate blood collection by venipuncture or have a history of fainting during acupuncture and seeing blood;

     20. Hepatitis B virus surface antigen (HbsAg) positive, or hepatitis C virus (HCV) antibody positive, or human immunodeficiency virus (HIV) antibody or Treponema pallidum antibody (TP-Ab) positive at screening;

     21. A history of alcohol abuse (drinking more than 14 units of alcohol per week [1 unit = 360 mL of beer with 5% alcohol, or 45 mL of spirits with 40% alcohol, or 150 mL of wine with 12% alcohol]) within 3 months prior to screening, subjects who have a positive alcohol breathalyzer test at baseline, or who are unable to abstain from alcohol during the study;

     22. History of drug abuse within 3 months prior to screening or a positive drug abuse screening (urine screen);

     23. Subjects who smoke ≥ 5 cigarettes per day within the 3 months prior to screening or who are unable to abstain from smoking throughout the study;

     24. Significantly active or unstable major depression or other major psychiatric conditions or any history of suicide attempt within 2 years prior to screening;

     25. Pregnant or lactating women;

     26. Have other conditions that, in the judgment of the investigator, make participation in this study inappropriate.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2023-11-21 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-10-17 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of a multiple escalation dose of ZT002 through the incidence and severity of treatment emergent adverse events in MAD Cohorts. Number of participants with treatment-emergent adverse events. | up to 270 days
Safety and tolerability of a multiple escalation dose of ZT002 through the incidence severity of serious adverse events in MAD Cohorts. Number of participants with serious adverse events. | up to 270 days

SECONDARY OUTCOMES:
The Pharmacokinetics (PK) profile of a multiple escalation dose of ZT002 in participants with overweight or obesity. | up to 270 days
  Parameter: Maximum observed plasma concentration of ZT002 (Css_max)
The Pharmacokinetics (PK) profile of a single escalation dose of ZT002 in participants with overweight or obesity. | up to 270 days
  Parameter: Area under the drug-time curve from 0 h after dosing to the last quantifiable concentration time point (AUC0-τ,SS)
The anti-drug antibody (ADA) response through testing serum or plasma of the participants post-dosing. | up to 270 days

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoli Li, Master, Principal Investigator — First Affiliated Hospital of Bengbu Medical College; Huan Zhou, PhD, Principal Investigator — First Affiliated Hospital of Bengbu Medical College
Locations (1):
- First Affiliated Hospital of Bengbu Medical College, Bengbu, China